CLINICAL TRIAL: NCT06400329
Title: Evaluating the Physiological Impact of Pain Neuroscience Education Versus Standard Education for Older Adults With Osteoarthritis
Brief Title: Physiological Impact of Different Types of Osteoarthritis Education.
Acronym: PNE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Carlesso (Other)
Responsible Party: Sponsor-Investigator, Lisa Carlesso, Associate Professor, PT PhD, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HiREB-16902
Record Dates: First submitted 2024-04-25; First posted 2024-05-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis; Chronic Pain
Keywords: Pain Neuroscience Education (PNE); Osteoarthritis; Autonomic Nervous System (ANS); Physiological responses; Biomedical education
MeSH Terms: conditions — Osteoarthritis; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to study hypotheses and the two treatment groups. As both arms of the study are providing education-based interventions, participants will be provided limited details of each intervention arm so as to blind them from knowing which is the intervention and which is the control. This will help minimize any bias that occurs by knowledge of group assignment and perception of treatment effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education (Experimental): The educational content will be presented to the participants at a computer station in the format of a website to navigate to simulate the experience and information that they may come across while browsing the internet for information about knee OA. The content will include 4 components, regardless of the education type. These components include knee osteoarthritis (OA)-related images, facts and myths, disease related concepts, and patient-doctor statements. The distinction between the two educational approaches lies in how information is presented. PNE focuses more on the neurophysiology of pain and approaches it from the perspective that knee OA pain is manageable, using neutral to positive language and emphasizes the importance of physical function and staying active. After the educational content is delivered, the participants will be shown the content again and will be asked to talk aloud about each page that they were shown.
  Interventions: Other: Pain Neuroscience Education
- Biomedical education (Active Comparator): In Standard Pain Education, the emphasis is on the structural pathology of knee OA and the outdated but common understanding of the disease process as a degenerative one, potentially conveying negative and threatening language.
  After the educational content is delivered, the participants will be shown the content again and will be asked to talk aloud about each page that they were shown.
  Interventions: Other: Standard Pain Education

INTERVENTIONS:
Other: Pain Neuroscience Education — PNE focuses more on the neurophysiology of pain and approaches it from the perspective that knee OA pain is manageable, using neutral to positive language and emphasizes the importance of physical function and staying active
  Arms: Pain neuroscience education
Other: Standard Pain Education — In Standard Pain Education, the emphasis is on the structural pathology of knee OA and the outdated but common understanding of the disease process as a degenerative one, potentially conveying negative and threatening language
  Arms: Biomedical education

SUMMARY:
In this study, the investigators are comparing two types of education for older adults with knee osteoarthritis: standard biomedical education focusing on the disease process, and a newer approach called pain neuroscience education (PNE), which teaches about the complexity of pain and dispels myths. While PNE has shown benefits in self-reported pain and function, little is known about its effects on physiological responses to pain.

the investigators will measure physiological indicators, particularly activity in the autonomic nervous system (ANS), which is closely linked to pain. Dysregulation in the ANS is common in chronic pain conditions like osteoarthritis. Our study aims to assess the feasibility of comparing these education methods and explore differences in physiological responses, as well as self-reported outcomes like cognitive and emotional factors.

Our goals are to determine if the study protocol is feasible, assess participants' acceptance of the assessment procedures, and explore differences in physiological markers and self-reported outcomes between the two education groups. Ultimately, the investigators aim to understand how different educational approaches may affect nervous system processing in older adults with knee osteoarthritis. the investigators hypothesize that those receiving PNE will show less autonomic arousal and nervous system sensitivity compared to those receiving standard education.

DETAILED DESCRIPTION:
Education and understanding of musculoskeletal (MSK) pain is known to be important for individuals and can improve patient outcomes (i.e. pain and function)(1). Many years ago, it became apparent that there was a vast disconnect between the scientific understanding of pain (i.e. its protective function, its complexity, and the most effective ways of treating it) and the current understanding of 'how pain works' held by patients and health professionals alike(2), one that was entrenched in an outdated biomedical model. Traditionally education has focused on the disease process which can have a negative impact with its language and images due to its focus on structural pathology.(3) Additionally, despite the known benefits of certain interventions e.g. exercise for MSK disorders, people may be wrongly advised that too much exercise could cause joint pain and damage.(4) Many of these poorly construed messages are due to a lack of understanding of the impact of such language, the complexity of the pain experience, and its lack of correlation with what the investigators now consider to be normal age-related changes seen on imaging.(2) The aim of intensive education about pain neuroscience was to give credibility to the best treatments available - active, psychological and self-management skills by providing a modern understanding of how pain works with the hope of giving power and agency to individuals to make optimal decisions about how to manage their health situation. Simply put, PNE aimed to enable and empower patients to adopt a biopsychosocial understanding of their problem and thereby pursue a biopsychosocial-based approach to overcoming it.(2) PNE involves the process of educating individuals about the complexity of pain and how our bodies process pain. It also seeks to dispel many of the myths long held by the public regarding MSK disorders(5). Despite PNE showing consistent positive effects on self-reported pain and function, there has been a growing debate in the literature regarding its value(6,7) Interestingly, there has been little to no evaluation of how differing approaches to education impacts people's physiological reactions and nervous system processing of pain. This project will fill that gap by providing unique understanding of how the type of educational content provided to older adults with knee osteoarthritis may impact their nervous system functioning and processing of pain.

Measuring pain remains a challenge, especially from a psycho-physiological aspect(8). Among various physiological indicators, the activity of the autonomic nervous system (ANS), specifically its sympathetic and parasympathetic subdivisions, is closely associated with pain (9). Enhanced activity in the sympathetic nervous system leads to increased electrodermal activity (sweating), respiration rate, heart rate, blood pressure, vascular vasoconstriction, and pupil dilation. In states of chronic pain, the autonomic nervous system may experience dysregulation, often resulting in diminished autonomic responsiveness to painful or stressful stimuli. Autonomic dysfunction has been observed in various chronic conditions, including knee osteoarthritis(10), low back pain(9), rheumatoid arthritis(11), and fibromyalgia(12). Targeting the dysregulated autonomic nervous system could potentially restore balance to stress response systems and alleviate systemic inflammation. The purpose of this pilot study will be to evaluate 1) the feasibility of a study protocol to investigate if there are differences in physiological responses associated with exposure to different types of knee osteoarthritis educational content. 2) to explore differences in the physiological responses between exposure to pain neuroscience education and standard biomedical education and 3) to explore differences in self-reported cognitive, emotional and functional outcomes and the physiological responses in each intervention arm

ELIGIBILITY:
Inclusion Criteria:

* ≥ 55-85years old
* community dwelling adults with a diagnosis of knee osteoarthritis or fulfilling the NICE criteria for knee OA
* activity-related joint pain
* either no morning joint-related stiffness or morning stiffness that lasts no longer than 30 minutes

Exclusion Criteria:

* those who have received prior PNE
* those who have eye glasses prescription exceeding +/- 6 for spherical correction and/or +3 for astigmatism

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Burden of the assessments | 1 week post-intervention
  Burden of completing the physical tests and questionnaires (0 = no burden, 10 = most burden)
feasibility outcomes (recruitment rate) | at 3 months
  36 participants consent to participate in 3 months; ≥24 participants consent to participate in 3 months; <24 participants consent to participate in 3 months
Feasibility outcomes (Educational content and format acceptability) | 1 week post-intervention
  ≥50% found content acceptable (Likert ≥4/5); ≥25% found content acceptable (Likert ≥4/5); <25% found content acceptable (Likert ≥4/5)
Feasibility outcomes (Lab Site accessibility/ Participant Convenience) | 1 week post-intervention
  ≥80% of participants find the lab accessible and convenient; ≥50% of participants find the lab accessible and convenient; <50% of participants find the lab accessible and convenient.
Feasibility outcomes (Scheduling of Lab assessments) | 1 week post-intervention
  ≥90% of scheduled assessments were on time; ≥75% of scheduled assessments were on time; >50% of scheduled assessments were on time.

SECONDARY OUTCOMES:
Demographic information | At baseline
  age, sex, gender, education, marital status, race, height, and weight
Temporal Summation (TS) | Before and after the delivery of the intervention
  Quantitative sensory testing in the form of mechanical temporal summation will be conducted to assess central nervous system sensitivity. We will use a 512mN weighted probe applied at the volar wrist opposite to the index knee (or least painful knee). It will be applied once and participants will be asked to rate their pain between 0 and 100.(16,17) Then, the same stimulus is applied 10 times at the rate of 1 per second and they are asked again to rate their pain. TS is defined as being present when, compared with the initial trial, the participant reports increased pain following the second trial.(16) This method has been used in many patient populations(18) including people with knee OA.(19)
Eye Tracker | During the delivery of the intervention
  Participants will be seated 63-65cm away from the display, which is the optimal distance determined by Tobii. Participants will be asked to fixate and follow with their gaze a red circle moving on the screen. The Tobii X2-60 Eye Tracker is an unobtrusive eye tracker for detailed research of natural eye gaze behavior. It is a standalone remote device (no contact with the participant) that is attached to the display. The tracker uses infrared diodes or LEDs to generate reflection patterns on the corneas of the participants' eyes. These reflection patterns, together with other visual data about the participants, are collected by the device's image sensors (at 60 Hz, or data points per second), and allows it to accurately calculate the participants' gaze point with high temporal and spatial precision. Its large head movement box allows the subject to move during recording while maintaining accuracy and precision.
Galvanic Skin Response | Before and during the delivery of the intervention
  Reciprocal of the measure of how much resistance the skin of an organism in a state of rest or basal activity offers to passage of an electrical current. For each participant only 2 electrodes are required at either of the locations indicated in the graphic. We will only be using locations 1-4 or 9-10 depending on which provides the best signal to noise ratio for each experimental task after pilot testing. Used with EL507 disposable snap electrodes that are designed for electrodermal activity studies and are pre-gelled with isotonic gel. The latex-free electrodes conform and adhere well to the body. The conductive gel used is medically approved BIOPAC non-irritating, isotonic Gel 101. It has the following components: Cetyl Alcohol #697313, Glycerol Monostearate, Lanolin, USP Anhydrous, Dimenthicon Silicone TBF9-1000, Water, purified USP Sodium Chloride, Sodium Lauryl Sulfate, Sorbitol, 70 USP, Methylparaben, Propylparaben, Quaternium-15
Heart Rate variability | Before and during delivery of the intervention
  ECG data will be collected with participants in a seated position to minimize potential parasympathetic saturation. Participants will be instructed to maintain regular sleep, avoid alcohol, and physical exercise within 24 hours of the visit. Participants will also empty their bladders before the session. Data acquisition will be performed using BIOPAC MP160 equipment. Participants will be instructed to remain motionless and silence throughout this period. Lead II will be chosen for data recording due to its anticipated higher R peak compared to leads I and III. Electrode placement will involve connecting the positive terminal to the lower left rib, the negative terminal to the right clavicle and grounding to the lower right rib. Heart Rate Variability (HRV) will be assessed using the Acqknowledge software, which is attached to the BioPac system (MP160, USA).
Respiratory Rate | Before and during delivery of the intervention
  To monitor respiration, a strain gauge respiration belt (BIOPAC SS5LB; BIOPAC Systems Inc., Coletta, CA, USA) will be positioned at the midpoint between the navel and xiphoid process. The acquired respiration rate data from the belt will be transmitted to the acquisition system and analyzed using AcqKnowledge software version 5.0.
  A small training task will be utilized to familiarize the participants with the experimental procedure, get them comfortable with the lab environment and to establish a baseline for each participant. Participants will be given instructions for the task, the outcome of this task will have no effect on the study findings.
Chronic pain self-efficacy | Before and after the delivery of the intervention
  The Self-Efficacy for Managing Chronic Disease 6-item scale (SEMCD-6) will be used to measure self-efficacy for chronic pain sufferers, with higher reported scores indicating higher self-efficacy.(21) Items are measured on a 0-10 scale with higher scores indicating higher self-efficacy. The SEMCD-6 has reported to have high internal consistency (Chronbach alpha of 0.88), sensitive to change, with significant correlations with other health outcomes.(22)
Anxiety symptoms | Before and after the delivery of the intervention
  The anxiety sub-scale of the Hospital Anxiety and Depression Scale (HADS) will be used to assess anxiety.(23) The HADS consists of 7 questions to measure anxiety with higher scores representing increased severity in anxiety symptoms. Each item is rated on a 4-point scale (ranging from 0 = no not at all, to 3 = yes definitely), for a total score ranging from 0-21. Two items are reverse scored (ranging from 3 = no not at all, to 0 = yes definitely). It is a brief and reliable measure of emotional distress in general in chronic populations including chronic pain and rheumatology.(24) Average sensitivity and specificity is ≥ 0.80.(24)
Fear of movement | Before and after the delivery of the intervention
  The Brief Fear of Movement Scale for Osteoarthritis (BFMSO) will be used to assess activity avoidance of participants due to pain-related fear of movement.(25) The BFMSO has 6 items that are derived from the Tampa Scale for Kinesiophobia (TSK) and uses a 4-point Likert scale with higher values indicating higher levels of kinesiophobia.(25) The BFMSO has adequate convergent validity with measures of pain (β=.30 to .41), physical functioning (β=.44 to .48), and psychological functioning (β=.36 to .37).(25)
Knee injury and outcomes | Before and after the delivery of the intervention
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, used to assess self-reported opinions about patients' knee and associated problems, while evaluating short-term and long-term consequences of knee injury. There are 42 items in 5 scored sub scales, of which two will be used: 1) pain, and 2) function in daily living (ADL). Scores range from 0-100 with zero representing extreme knee problems and 100 representing no knee problems.(26) KOOS has adequate internal consistency (0.70-0.95) and construct validity in adults with knee OA.(27) Multiple studies have determined convergent and divergent construct validity with comparison to several instruments including the subscales of SF-36 and the Lysholm knee scoring scale.(28)
eHEALS | Before the delivery of the intervention
  Electronic health literacy was defined initially as "the ability to seek, find, understand, and appraise health information from electronic sources and apply the knowledge gained to addressing or solving a health problem" (p.2)(29). One of the measures of electronic health literacy is eHEALS. It comprises 8 items and respondents rate each item on a 5-point Likert Scale spanning from 1 (strongly disagree) to 5 (strongly agree). The higher value in each item represents a greater perception of eHealth literacy (30). eHEALS has adequate internal consistency (α = .94) and validity in adults with knee OA(31).
The Osteoarthritis Conceptualization Questionnaire | Before and after the delivery of the intervention
  The Osteoarthritis Conceptualization Questionnaire (OACQ) aims to explore individuals' perspectives on osteoarthritis and physical activity through a set of statements. Respondents are instructed to express their agreement or disagreement on a scale ranging from "Strongly Disagree=1" to "Strongly Agree=5." The questionnaire is divided into four sections: Influence of Variables, Physiology, Expectations, and Conceptual Change. Each section involves specific items, and some require reverse scoring. The OACQ demonstrates good test-retest reliability (ICC(3,1)= 0.89). Measures of convergent validity revealed a moderate correlation with other related scales.
The Intention to Exercise scale | Before and after the delivery of the intervention
  The Intention to Exercise scale involves three key questions: "I am committed to engage in physical activity over the next 2 weeks"; "I am motivated to engage in physical activity over the next 2 weeks" and "I am determined to engage in physical activity over the next 2 weeks"(32) . Participants are asked to rate their agreement on a 7-point Likert scale, ranging from "very strongly disagree" to "very strongly agree," This scale offers an understanding of participants' intentions and attitudes towards incorporating physical activity into their lives(33).
The surgery intention scale | Before and after the delivery of the intervention
  The surgery intention scale aimed to assess individuals' inclination toward knee joint replacement surgery. The responses, ranging from 'Yes,' 'No,' to 'Unsure,' provide valuable data on immediate surgery acceptance. This scale offers a comprehensive understanding of participants' attitudes and intentions regarding this specific surgical intervention (6).
The Self-Administered Comorbidity Questionnaire (SCQ) | Before the delivery of the intervention
  The self-administered comorbidity questionnaire (SCQ) is a highly effective tool for evaluating comorbid conditions in both clinical and health services research. The SCQ is brief, easy to understand, and can be completed by individuals without a medical background. It allows patients to indicate the severity of each comorbid condition and how it affects their daily functioning. The questionnaire includes 12 specific medical problems and 3 optional conditions. The SCQ shows modest correlations with a commonly used medical record-based comorbidity tool and with future health status and utilization.
Satisfaction with Information Quality | After the delivery of the intervention
  Satisfaction with information quality aims to capture respondents' views regarding the overall quality of information on a website using a 7-point Likert scale. Participants are prompted to assess their satisfaction levels across four dimensions: "Very dissatisfied" to "Very satisfied" (IQ1), "Very displeased" to "Very pleased" (IQ2), "Frustrated" to "Contented" (IQ3), and "Disappointed" to "Delighted" (IQ4). This comprehensive approach enables an understanding of users' perspectives on the quality of information available. This questionnaire demonstrated Adequate reliability. (Cronbach alpha>0.97)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carlesso, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Moseley L. Unraveling the barriers to reconceptualization of the problem in chronic pain: the actual and perceived ability of patients and health professionals to understand the neurophysiology. J Pain. 2003 May;4(4):184-9. doi: 10.1016/s1526-5900(03)00488-7. PMID 14622702
- [Background] Domenech J, Sanchez-Zuriaga D, Segura-Orti E, Espejo-Tort B, Lison JF. Impact of biomedical and biopsychosocial training sessions on the attitudes, beliefs, and recommendations of health care providers about low back pain: a randomised clinical trial. Pain. 2011 Nov;152(11):2557-2563. doi: 10.1016/j.pain.2011.07.023. Epub 2011 Sep 13. PMID 21917377
- [Background] Nissen N, Holm PM, Bricca A, Dideriksen M, Tang LH, Skou ST. Clinicians' beliefs and attitudes to physical activity and exercise therapy as treatment for knee and/or hip osteoarthritis: a scoping review. Osteoarthritis Cartilage. 2022 Feb;30(2):260-269. doi: 10.1016/j.joca.2021.11.008. Epub 2021 Nov 17. PMID 34800632
- [Background] Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. J Pain. 2015 Sep;16(9):807-13. doi: 10.1016/j.jpain.2015.05.005. Epub 2015 Jun 5. PMID 26051220
- [Background] Bonatesta L, Ruiz-Cardenas JD, Fernandez-Azorin L, Rodriguez-Juan JJ. Pain Science Education Plus Exercise Therapy in Chronic Nonspecific Spinal Pain: A Systematic Review and Meta-analyses of Randomized Clinical Trials. J Pain. 2022 Apr;23(4):535-546. doi: 10.1016/j.jpain.2021.09.006. Epub 2021 Oct 20. PMID 34678468
- [Background] Ordonez-Mora LT, Morales-Osorio MA, Rosero ID. Effectiveness of Interventions Based on Pain Neuroscience Education on Pain and Psychosocial Variables for Osteoarthritis: A Systematic Review. Int J Environ Res Public Health. 2022 Feb 23;19(5):2559. doi: 10.3390/ijerph19052559. PMID 35270250
- [Background] Otis JD. Flor, H., & Turk, D. C. (2011)Chronic Pain: An Integrated Biobehavioral Approach Seattle: IASP Press. Cogn Behav Pract. 2013 Feb 1;20(1):117-8.
- [Background] El-Badawy MA, El Mikkawy DM. Sympathetic Dysfunction in Patients With Chronic Low Back Pain and Failed Back Surgery Syndrome. Clin J Pain. 2016 Mar;32(3):226-31. doi: 10.1097/AJP.0000000000000250. PMID 25968450
- [Background] Bossenger NR, Lewis GN, Rice DA, Shepherd D. The autonomic and nociceptive response to acute exercise is impaired in people with knee osteoarthritis. Neurobiol Pain. 2023 Jan 19;13:100118. doi: 10.1016/j.ynpai.2023.100118. eCollection 2023 Jan-Jul. PMID 36711216
- [Background] Adlan AM, Paton JF, Lip GY, Kitas GD, Fisher JP. Increased sympathetic nerve activity and reduced cardiac baroreflex sensitivity in rheumatoid arthritis. J Physiol. 2017 Feb 1;595(3):967-981. doi: 10.1113/JP272944. Epub 2016 Oct 24. PMID 27561790
- [Background] Reyes del Paso GA, Garrido S, Pulgar A, Duschek S. Autonomic cardiovascular control and responses to experimental pain stimulation in fibromyalgia syndrome. J Psychosom Res. 2011 Feb;70(2):125-34. doi: 10.1016/j.jpsychores.2010.09.012. Epub 2010 Nov 18. PMID 21262414
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] NICE [Internet]. NICE; [cited 2024 Jan 29]. Osteoarthritis | NICE impact arthritis | Reviewing the impact of our guidance | Measuring the use of NICE guidance | Into practice | What we do | About. Available from: https://www.nice.org.uk/about/what-we-do/into-practice/measuring-the-use-of-nice-guidance/impact-of-our-guidance/nice-impact-arthritis/osteoarthritis
- [Background] Neogi T, Frey-Law L, Scholz J, Niu J, Arendt-Nielsen L, Woolf C, Nevitt M, Bradley L, Felson DT; Multicenter Osteoarthritis (MOST) Study. Sensitivity and sensitisation in relation to pain severity in knee osteoarthritis: trait or state? Ann Rheum Dis. 2015 Apr;74(4):682-8. doi: 10.1136/annrheumdis-2013-204191. Epub 2013 Dec 18. PMID 24351516
- [Background] Neogi T, Guermazi A, Roemer F, Nevitt MC, Scholz J, Arendt-Nielsen L, Woolf C, Niu J, Bradley LA, Quinn E, Law LF. Association of Joint Inflammation With Pain Sensitization in Knee Osteoarthritis: The Multicenter Osteoarthritis Study. Arthritis Rheumatol. 2016 Mar;68(3):654-61. doi: 10.1002/art.39488. PMID 26554395
- [Background] Plews DJ, Laursen PB, Stanley J, Kilding AE, Buchheit M. Training adaptation and heart rate variability in elite endurance athletes: opening the door to effective monitoring. Sports Med. 2013 Sep;43(9):773-81. doi: 10.1007/s40279-013-0071-8. PMID 23852425
- [Background] Yarnitsky D, Granot M, Nahman-Averbuch H, Khamaisi M, Granovsky Y. Conditioned pain modulation predicts duloxetine efficacy in painful diabetic neuropathy. Pain. 2012 Jun;153(6):1193-1198. doi: 10.1016/j.pain.2012.02.021. Epub 2012 Apr 3. PMID 22480803
- [Background] Finan PH, Buenaver LF, Bounds SC, Hussain S, Park RJ, Haque UJ, Campbell CM, Haythornthwaite JA, Edwards RR, Smith MT. Discordance between pain and radiographic severity in knee osteoarthritis: findings from quantitative sensory testing of central sensitization. Arthritis Rheum. 2013 Feb;65(2):363-72. doi: 10.1002/art.34646. PMID 22961435
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. J Clin Epidemiol. 2014 Nov;67(11):1265-73. doi: 10.1016/j.jclinepi.2014.06.009. Epub 2014 Aug 3. PMID 25091546
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Smarr KL, Keefer AL. Measures of depression and depressive symptoms: Beck Depression Inventory-II (BDI-II), Center for Epidemiologic Studies Depression Scale (CES-D), Geriatric Depression Scale (GDS), Hospital Anxiety and Depression Scale (HADS), and Patient Health Questionnaire-9 (PHQ-9). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S454-66. doi: 10.1002/acr.20556. No abstract available. PMID 22588766
- [Background] Shelby RA, Somers TJ, Keefe FJ, DeVellis BM, Patterson C, Renner JB, Jordan JM. Brief Fear of Movement Scale for osteoarthritis. Arthritis Care Res (Hoboken). 2012 Jun;64(6):862-71. doi: 10.1002/acr.21626. Epub 2012 Jan 30. PMID 22290689
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Collins NJ, Prinsen CA, Christensen R, Bartels EM, Terwee CB, Roos EM. Knee Injury and Osteoarthritis Outcome Score (KOOS): systematic review and meta-analysis of measurement properties. Osteoarthritis Cartilage. 2016 Aug;24(8):1317-29. doi: 10.1016/j.joca.2016.03.010. Epub 2016 Mar 21. PMID 27012756
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746
- [Background] Norman CD, Skinner HA. eHealth Literacy: Essential Skills for Consumer Health in a Networked World. J Med Internet Res. 2006 Jun 16;8(2):e9. doi: 10.2196/jmir.8.2.e9. PMID 16867972
- [Background] Chung SY, Nahm ES. Testing reliability and validity of the eHealth Literacy Scale (eHEALS) for older adults recruited online. Comput Inform Nurs. 2015 Apr;33(4):150-6. doi: 10.1097/CIN.0000000000000146. PMID 25783223
- [Background] Rhodes RE, Hunt Matheson D, Mark R. Evaluation of Social Cognitive Scaling Response Options in the Physical Activity Domain. Meas Phys Educ Exerc Sci. 2010 Jul 30;14(3):137-50.
- [Background] Stanton TR, Braithwaite FA, Butler D, Moseley GL, Hill C, Milte R, Ratcliffe J, Maher C, Tomkins-Lane C, Pulling BW, MacIntyre E, Esterman A, Stanford T, Lee H, Fraysse F, Metcalf B, Mouatt B, Bennell K. The EPIPHA-KNEE trial: Explaining Pain to target unhelpful pain beliefs to Increase PHysical Activity in KNEE osteoarthritis - a protocol for a multicentre, randomised controlled trial with clinical- and cost-effectiveness analysis. BMC Musculoskelet Disord. 2021 Aug 28;22(1):738. doi: 10.1186/s12891-021-04561-6. PMID 34454458